CLINICAL TRIAL: NCT03426618
Title: A Real-World Observational Study for the Safety and Efficacy of Baraclude (Entecavir) in Korean Pediatric (Aged 2-16 Years) Patients With Chronic Hepatitis B
Brief Title: A Real-World Observational Study for the Safety and Efficacy of Baraclude in Korean Pediatric Patients With Chronic Hepatitis B
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: AI463-514
Record Dates: First submitted 2018-02-02; First posted 2018-02-08 (Actual); Last update posted 2019-06-03 (Actual); Status verified 2019-05

CONDITIONS: Hepatitis B
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pediatric participants with Hepatitis B Virus (HBV): All participants who received at least 1 dose of Baraclude.
  Interventions: Other: Non-interventional

INTERVENTIONS:
Other: Non-interventional — Non-interventional

SUMMARY:
This is a local, prospective observational study (regulatory post marketing surveillance) to access the safety and effectiveness of Baraclude in Korean pediatric patients with chronic HBV infection who are between the ages of 2 and less than 16 years.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* 2 to < 16 years of age
* Patients with chronic hepatitis B infection, eligible for treatment with Baraclude as indicated in the locally approved prescribing information

Exclusion Criteria:

* Off-label use of the approved label in Baraclude pediatric indication
* Patients with a contraindication for the use of Baraclude as described in the locally approved prescribing information

Other protocol defined inclusion/exclusion criteria could apply

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Participants will be enrolled with chronic hepatitis B virus (CHB)between the ages of 2 and less than 16 years and who will begin treatment with Baraclude.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2018-01-12 (Actual); Primary Completion 2019-03-13 (Actual); Study Completion 2019-03-13 (Actual)

PRIMARY OUTCOMES:
Number of Adverse Events (AEs) | Up to 52 weeks

SECONDARY OUTCOMES:
Participants who achieved a virologic response | Up to 48 weeks
  Measured by reduction in hepatitis B virus DNA to <300 copies/mL
Mean log reduction in hepititis B virus DNA | Baseline to Weeks 12, 24, and 48
Liver stiffness | Baseline and Week 48 of treatment
Number of participants with resistance to Baraclude | Up to 52 weeks
Number of participants with virologic relapse in participants | Up to 48 weeks
  Viral load of less than or equal to 300 copies/mL
Number of participants with virologic Relapse in participants | Up to 48 weeks
  Viral load greater than 10,000 copies/mL
Number of participants who were HBeAg seroconverted at Week 48 | Week 48
Number of participants who had HBeAg loss at week 48 | Week 48
Number of participants who were HBsAg seroconverted at Week 48 | Week 48
Number of participants who had HBsAg loss at week 48 | Week 48
Number of participants with normalization of serum ALT at week 12 | Baseline to week 12
  Normalization is measured as less than or equal to 1 X the upper limit of normal of serum ALT
Number of participants with normalization of serum ALT at week 24 | Baseline to week 24
  Normalization is measured as less than or equal to 1 X the upper limit of normal of serum ALT
Number of participants with normalization of serum ALT at week 48 | Baseline to week 48
  Normalization is measured as less than or equal to 1 X the upper limit of normal of serum ALT

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Seoul, South Korea

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm